CLINICAL TRIAL: NCT03517644
Title: Hope and Expectations as Components of Open-Label Placebos: An Experimental Study Investigating Pain
Brief Title: Investigating Hope and Expectations in Open-Label Placebos
Acronym: I-HELP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-58v
Record Dates: First submitted 2018-03-07; First posted 2018-05-07 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of four experimental groups in parallel for the duration of the study
Who Masked: Participant
Masking Description: Using a cover story, participants are instructed to think that there are three experimental groups: a treatment condition, a placebo condition, and a control condition. Therefore, participants from the open-label groups do know that they receive a placebo, but do not know which specific mechanism is being addressed in their condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Deceptive Placebo (DP) (Experimental): After pretreatment heat pain assessment, participants are informed that they are about to receive an effective analgesic cream. In fact, they receive a placebo cream. Next, the posttreatment pain assessment is conducted.
  Interventions: Other: DP; Other: Placebo cream; Other: Heat pain
- OLP with Hope (OLP Hope) (Experimental): After pretreatment heat pain assessment, participants are informed that they are about to receive an placebo cream. They are told that the cream has no active pharmacological ingredient. However, using verbal instructions, the investigator aims to induce hope among the participants that the cream could have a positive effect. Next, the posttreatment pain assessment is conducted.
  Interventions: Other: OLP Hope; Other: Placebo cream; Other: Heat pain
- OLP with Expectations (OLP Expectation) (Experimental): After pretreatment heat pain assessment, participants are informed that they are about to receive an placebo cream. They are told that the cream has no active pharmacological ingredient. However, using verbal instructions, the investigator aims to raise expectations among the participants that the cream will have a positive effect. Next, the posttreatment pain assessment is conducted.
  Interventions: Other: OLP Expectation; Other: Placebo cream; Other: Heat pain
- Control (Experimental): After pretreatment heat pain assessment, this group does not receive an intervention targeting pain sensation prior to the posttreatment pain assessment.
  Interventions: Other: Heat pain

INTERVENTIONS:
Other: DP — Participants are informed that they are about to receive an effective analgesic cream. They are instructed to apply the cream using a cotton pad.
  Arms: Deceptive Placebo (DP)
Other: OLP Hope — Participants are informed that they are about to receive an placebo cream. They are told that the cream has no active pharmacological ingredient. Therefore, participants are supposed to evaluate the subjective probability for a positive effect of the cream as rather low. However, using verbal instructions, the investigator aims to induce hope among the participants that the cream could have a positive effect for them because this placebo cream did have a positive among some former participants who were similar to the current participant. The emphasis of this similarity (regarding age and sex) aims to induce a feeling of connectedness to previous participants who reported positive effects of the placebo cream.
  Arms: OLP with Hope (OLP Hope)
Other: OLP Expectation — Participants are informed that they are about to receive an placebo cream. They are told that the cream has no active pharmacological ingredient. However, participants are told that placebos have been shown to contribute substantially to clinical outcomes such as pain intensity/unpleasantness. This positive effect of placebos is reasoned by explaining learning mechanisms such as classical conditioning. We anticipated that after hearing this instruction, participants would consider it to be likely that the placebo has a positive effect for them.
  Arms: OLP with Expectations (OLP Expectation)
Other: Placebo cream — The participants receive an inert placebo cream (standard basic cream with oil of thyme produced by a local pharmacy).
  Arms: Deceptive Placebo (DP); OLP with Expectations (OLP Expectation); OLP with Hope (OLP Hope)
Other: Heat pain — Participant receive heat pain stimuli using the suprathreshold method of the Thermo Sensory Analyser (TSA-II), a commonly used device to study pain sensation and analgesic effects.

SUMMARY:
Research has shown that placebo effects contribute substantially to clinical outcomes. Recent evidence suggests that placebos remain effective even if they are openly described as placebos (so-called Open-Label Placebos). In this study, the investigators examine hope and expectations as components of open-label placebos in an experimental study investigating pain..

DETAILED DESCRIPTION:
A growing body of research has indicated that placebos contribute substantially to clinical outcomes. Yet, the implementation of deceptive placebos in clinical practice is incompatible with key principles of openness and patient autonomy. However, recent research suggests that placebos remain effective even if they openly described as placebos (so-called Open-Label Placebos (OLP)), hence questioning the necessity of deception in clinical trials. However, research identifying the specific mechanisms underlying OLP is lacking. Therefore, the current study aims to examine hope and expectations as components of OLP in pain.

For this purpose, experimentally induced heat pain is examined. First, all participants receive heat pain stimuli and evaluate them. Next, participants are randomly assigned to one of four groups: (1) a traditional deceptive placebo (DP) group, which is told that they receive an effective analgesic cream, (2) an OLP group inducing hope among the participants that the placebo cream could help them tolerating painful stimuli (OLP hope), (3) and OLP group raising the expectation that the placebo cream will help participants tolerating heat pain (OLP expectation), (4) a control group receiving no cream. Finally, participants receive and evaluate heat pain again.

ELIGIBILITY:
Inclusion Criteria:

* sufficient German language knowledge
* at least 18 years old

Exclusion Criteria:

* current mental disorder
* current medical disease
* studying psychology or medicine
* pregnancy or breastfeeding period
* intake of drugs
* severely visually impaired

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-02-10 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-08-21 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity scale | Baseline and 45 minutes
  Change in subjective pain intensity assessed using a visual analogue scale (ranging from 0 to 100, with higher values reflecting more pain intensity)

SECONDARY OUTCOMES:
Change in pain unpleasantness scale | Baseline and 45 minutes
  Change in subjective pain unpleasantness assessed using a visual analogue scale (ranging from 0 to 100, with higher values reflecting more pain unpleasantness)
Change in physiological heat pain threshold | Baseline and 45 minutes
  Change in the individual heat pain threshold (the point when the stimulus changes from being warm to being painful)
Change in physiological heat pain tolerance | Baseline and 45 minutes
  Change in the individual heat pain tolerance (the point when participants cannot stand the heat pain stimulus any longer)

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Kube, M. Sc., Principal Investigator — Philipps University Marburg
Locations (1):
- Philipps-University of Marburg, Marburg, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared